CLINICAL TRIAL: NCT02595242
Title: Safety and Efficacy Study of Mitoxantrone Hydrochloride Liposome Injection Plus Cyclophosphamide,Vincristine and Prednison (CNOP)in Diffuse Large B Cell Lymphoma
Brief Title: Safety and Efficacy Study of CNOP Chemotherapy in Diffuse Large B Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-HE1505/PRO/Ⅰ
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mitoxantrone 12 mg/m2 (Experimental): Mitoxantrone Hydrochloride Liposome Injection 12 mg/m2 will be infused intravenously once over 1 hours in 250 ml 5％ glucose injection on the first day during a treatment phase of 3 weeks.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone
- Mitoxantrone 16 mg/m2 (Experimental): Mitoxantrone Hydrochloride Liposome Injection 16 mg/m2 will be infused intravenously once over 1 hours in 250 ml 5％ glucose injection on the first day during a treatment phase of 3 weeks.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone
- Mitoxantrone 20mg/m2 (Experimental): Mitoxantrone Hydrochloride Liposome Injection 20 mg/m2 will be infused intravenously once over 1 hours in 250 ml 5％ glucose injection on the first day during a treatment phase of 3 weeks.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 will be infused intravenously once 1-2 minutes in 20-30 ml saline on the first day during a treatment phase of 3 weeks.
Drug: Vincristine — Vincristine 0.3-0.5 mg/ml will be infused intravenously once about 5 minutes in saline on the first day during a treatment phase of 3 weeks.
Drug: Prednisone — Prednisone 100 mg/d will be taken orally on the first 1-5 day during a treatment phase of 3 weeks.

SUMMARY:
The purpose of this study is to determine whether Mitoxantrone Hydrochloride Liposome Injection plus Cyclophosphamide,Vincristine and Prednison(CNOP)is safe and effective in the treatment of Diffuse Large B Cell Lymphoma.

DETAILED DESCRIPTION:
Mitoxantrone Hydrochloride Liposome Injection is a kind of anthraquinone compounds, and its antineoplastic effect has been viewed in preclinical tests. The investigator´s phaseⅠstudy has shown that the drug´s toxicity is manageable and the tolerable does is 20 mg/m2. The purpose of this study is to determine whether Mitoxantrone Hydrochloride Liposome Injection plus Cyclophosphamide,Vincristine and Prednison(CNOP)is safe and effective in the treatment of Diffuse Large B Cell Lymphoma.Patients physical state, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if Mitoxantrone Hydrochloride Liposome Injection plus Cyclophosphamide,Vincristine and Prednison(CNOP)is safe and effective in the treatment of Diffuse Large B Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to study specific screening procedures;
* Favorable index of curative effect of Diffuse Large B Cell Lymphoma confirmed by histological analysis;
* ≥ 18 and ≤ 70 years of age, male or female;
* Advanced Lymphoma and standard treatments failed;
* May benefit from anthracycline-based drugs;
* ECOG performance status of 0-2;
* More than 4 weeks from the last chemotherapy, more than 4 weeks from the last biotherapy, more than 4 weeks from the last clinical trial drug therapy;
* Life expectancy of more than 3 months;
* Sexually active women of childbearing potential must use a medically acceptable form of contraception;
* Adequate hepatic, renal, cardiac and hematologic functions: leukocyte≥3.5×10^9/L,neutrophils≥2.0×10^9/L,platelets≥100×10^9/L, hemoglobin≥90g/L,creatinine clearance rate≤1.5×ULN, serum bilirubin≤1.5×ULN, ALT≤2.5×ULN(5×for liver metastasis),AST≤2.5×ULN(5×for liver metastasis), alkaline phosphatase≤200 IU/L,Electrocardiogram appeared to be essentially normal, ejection fraction of Heart Doppler ultrasound appeared to be normal.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients with Multiple sclerosis;
* Suffering from serious internal disease, including serious heart attack, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension,uncontrolled infection, Active peptic ulcer;
* Mitoxantrone has been used before;
* The cumulative does of doxorubicin and epirubicin before inclusion have surpassed 360 mg/m2 and 600 mg/m2, respectively;
* Heart disease was caused after Anthracycline-based drugs used;
* Other antineoplastic drugs need to be used in this study;
* History of Anthracycline-based drug allergy or liposome drug allergy;
* Uncontrolled primary brain tumor or brain metastases;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective response rate) | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huaqing Wang, Ph.D, Principal Investigator — Tianjin People's Hospital
Locations (1):
- Tianjin people's Hospital, Tianjin, China